CLINICAL TRIAL: NCT05682443
Title: Randomized Study of ONC-392 Plus Lutetium Lu 177 Vipivotide Tetraxetan in Patients With Metastatic Castration-Resistant Prostate Cancer (mCRPC) Who Progressed on Androgen Receptor (AR) Pathway Inhibition
Brief Title: ONC-392 Plus Lutetium Lu 177 Vipivotide Tetraxetan in Patients With mCRPC
Acronym: PRESERVE-006
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: OncoC4, Inc. (Industry)
Collaborators: Prostate Cancer Clinical Trials Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRESERVE-006
Record Dates: First submitted 2022-12-26; First posted 2023-01-12 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
MeSH Terms: interventions — Pluvicto

STUDY DESIGN:
Intervention Model Description: Randomized, open label, active controlled, multi-center study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: ONC-392 low dose plus lutetium Lu 177 vipivotide tetraxetan (Experimental): Arm 1 receives ONC-392 3 mg/kg, IV infusion, Q4W for up to 13 doses, plus lutetium Lu 177 vipivotide tetraxetan IV infusion, Q6W for up to 6 doses.
  Interventions: Drug: ONC-392 low; Drug: lutetium Lu 177 vipivotide tetraxetan
- Arm 2: ONC-392 high dose plus lutetium Lu 177 vipivotide tetraxetan (Experimental): Arm 2 receives ONC-392 6 mg/kg, IV infusion, Q6W for up to 9 doses, plus lutetium Lu 177 vipivotide tetraxetan IV infusion, Q6W for up to 6 doses.
  Interventions: Drug: ONC-392 high; Drug: lutetium Lu 177 vipivotide tetraxetan
- Arm 3: lutetium Lu 177 vipivotide tetraxetan (Active Comparator): Arm 3 receives lutetium Lu 177 vipivotide tetraxetan, IV infusion, Q6W for up to 6 doses.
  Interventions: Drug: lutetium Lu 177 vipivotide tetraxetan

INTERVENTIONS:
Drug: ONC-392 low — ONC-392 will be given as IV infusion, Q4W for up to 13 doses.
  Other Names: A humanized anti-CTLA4 IgG1 monoclonal antibody; Gotistobart
  Arms: Arm 1: ONC-392 low dose plus lutetium Lu 177 vipivotide tetraxetan
Drug: ONC-392 high — ONC-392 will be given as IV infusion, Q6W for up to 9 doses.
  Other Names: A humanized anti-CTLA4 IgG1 monoclonal antibody; Gotistobart
  Arms: Arm 2: ONC-392 high dose plus lutetium Lu 177 vipivotide tetraxetan
Drug: lutetium Lu 177 vipivotide tetraxetan — lutetium Lu 177 vipivotide tetraxetan will be given as IV infusion, Q6W, for up to 6 doses.
  Other Names: Pluvicto

SUMMARY:
In this Phase 2 study, mCRPC patients with PSMA positive scans who progressed on prior ARTA and up to 2 lines of taxanes, and are naïve to lutetium Lu 177 vipivotide tetraxetan, will be enrolled. The study is open-label, randomized with active control, multi-center study.

DETAILED DESCRIPTION:
The goal of this clinical trial is to examine the safety and efficacy of ONC-392 in combination with lutetium Lu 177 vipivotide tetraxetan in metastatic castration resistant prostate cancer patient who have disease progressed on androgen receptor pathway inhibition. The main questions it aims to answer are (1) whether it is safe to combine ONC-392 with lutetium Lu 177 vipivotide tetraxetan, (2) whether the combination increases the radiographic progression free survival (rPFS).

In Phase 1 of the trial, participates will be randomized to experimental arm and control arm in 2:1 ratio. In experimental arm, they will be given ONC-392 IV infusion for up to 9 cycles or approximately one year, together with lutetium Lu 177 vipivotide tetraxetan for up to 6 cycles. In Phase 2 of the trial, participants will be randomized to three arms in 1:1:1 ratio. There will be two experimental arms, one with low dose of ONC-392 and one with high dose ONC-392, to be given in IV infusion for up to 9 or 13 cycles or approximately one year, together with lutetium Lu 177 vipivotide tetraxetan for up to 6 cycles. In active control arm for both Phase 1 and Phase 2, participants will be given standard of care treatment with lutetium Lu 177 vipivotide tetraxetan for up to 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be ≥ 18 years of age and have the ability to understand and sign an approved informed consent form (ICF).
2. Patients must have an ECOG performance status of 0 or 1.
3. Patients must have a life expectancy > 6 months.
4. Patients must have histological or cytological confirmation of prostate adenocarcinoma.
5. Patients must have a positive PSMA in an FDA-approved PSMA PET scan. A positive PSMA is defined as at least one tumor lesion with PSMA uptake greater than normal liver.
6. Patients must have prior orchiectomy and/or ongoing androgen-deprivation therapy and a castrate level of serum testosterone (< 50 ng/dL or < 1.7 nmol/L).
7. Patients must have received at least one second generation AR-targeting agents (such as apalutamide, darolutamide, enzalutamide and/or abiraterone).
8. Patients should have prior treatment of up to two taxane regimens, or are unfit for, or refuse taxane chemotherapy. A taxane regimen is defined as a minimum exposure of 2 cycles of a taxane. Note: Taxane chemotherapy administered in the Castration Sensitive Prostate Cancer (CSPC) or Castration Resistant Prostate Cancer (CRPC) setting is allowed.
9. Patients must have progressive mCRPC. Documented progressive mCRPC will be based on at least 1 of the following criteria:

   1. Serum PSA progression defined as 2 consecutive increases in PSA over a previous reference value measured at least 1 week prior. The minimal start value is 1.0 ng/mL.
   2. RECIST v1.1 soft-tissue progression
   3. Progression of bone disease: 2 or more new metastatic bone lesions by bone scan per PCWG3 criteria.
10. Patients must have ≥ 1 metastatic lesion that is present on baseline CT, MRI, or bone scan imaging obtained ≤ 42 days prior to beginning study therapy.
11. Patients must have adequate organ function.
12. Patients with or without concomitant bisphosphonate or denosumab regimen for ≥ 30 days prior to randomization are eligible.
13. For patients who have partners of childbearing potential: Partner and/or patient must use adequate methods of birth control with barrier protection, deemed acceptable by the principal investigator during the study and for 3 months after last study drug administration.

Exclusion Criteria:

1. Patients who have not recovered to NCI CTCAE grade ≤ 1 from an adverse event (AE) due to prior cancer therapeutics except neuropathy or endocrinopathy with Gr 2 or less.
2. Any systemic anti-cancer therapy within 5 half-lives or 14 days, whichever is shorter (small molecule drugs) or within 28 days for antibody based therapy, prior to starting study treatment.
3. Known hypersensitivity to the components of the study therapy or its analogs.
4. Other concurrent cytotoxic chemotherapy, immunotherapy, radioligand therapy, or investigational therapy.
5. Transfusion within 14 days of first day of study treatment
6. PSMA-negative lesions are defined as lesions with PSMA uptake equal to or lower than that of liver parenchyma. Patients with PSMA-negative lesions in any lymph node with a short axis of ≥ 2.5 cm, in any metastatic solid-organ lesions with a short axis of ≥ 1.0 cm, or in any metastatic bone lesion with a soft-tissue component of ≥ 1.0 cm in the short axis are ineligible.
7. Previous treatment with Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Radium-223 or hemi-body irradiation within 6 months prior to randomization. Previous PSMA-targeted radioligand therapy is not allowed.
8. Patients with a history of CNS metastases must have received therapy (surgery, radiotherapy, gamma knife) and be neurologically stable, asymptomatic, and not receiving corticosteroids for the purposes of maintaining neurologic integrity. Patients with epidural disease, canal disease and prior cord involvement are eligible if those areas have been treated, are stable, and not neurologically impaired. For patients with parenchymal CNS metastasis (or a history of CNS metastasis), baseline and subsequent radiological imaging must include evaluation of the brain (MRI preferred or CT with contrast).
9. A superscan as seen in the baseline bone scan.
10. Symptomatic cord compression, or clinical or radiologic findings indicative of impending cord compression.
11. Concurrent serious (as determined by the Principal Investigator) medical conditions, including, but not limited to, myocardial infarction within 6 months, New York Heart Association class III or IV congestive heart failure, history of congenital prolonged QT syndrome, or unstable arrhythmia within 3 months, uncontrolled infection, active hepatitis B or C, or other significant co-morbid conditions that in the opinion of the investigator would impair study participation or cooperation.
12. Active concurrent malignancy (with the exception of non-melanomatous skin cancer). Patients with carcinoma in situ of any origin and patients with prior malignancies who are in remission and/or whose likelihood of recurrence is very low per investigator's judgment are eligible for this study.
13. Receiving systemic steroid therapy with > 10 mg/day prednisone or equivalent within 7 days prior to the first dose of study treatment or receiving any other form of immunosuppressive medication.
14. Active GI disease, including peptic ulcer disease, pancreatitis, diverticulitis, or inflammatory bowel disease.
15. Active or previously documented autoimmune disease and/or current use of immunosuppressive agents. Use of endocrine replacement therapy (e.g., thyroxine, insulin, low dose of steroid, etc.) is allowed.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2023-12-11 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
PSA50 | 30 months
  Decrease in prostate-specific antigen (PSA) levels of at least 50% from baseline.
TEAEs and irAEs | 30 months
  Incidence of TEAEs, irAEs, and TEAEs leading to study treatment discontinuation.

SECONDARY OUTCOMES:
Composite radiographic progression-free survival (PFS) | 30 months
  Composite radiographic PFS by investigator. Disease progression as defined by PCWG3 guideline.
Composite progression-free survival (PFS) | 30 months
  The PFS event is defined as either radiographic progression, or PSA increase by PCWG3 guideline, or death, whichever comes first.
Overall survival (OS) | 30 months
  The length of time patients live after starting treatment.
Response rate | 30 months
  Response rate based on radiographic evaluation of PCWG3.
DoR (Duration of Response) and DCR (Disease Control Rate) | 30 months
  DoR and DCR based on radiographic evaluation of PCWG3. DoR and DCR based on PCWG3.

CONTACTS AND LOCATIONS:
Overall Officials: David Wise, MD, Principal Investigator — NYU Langone Health; Mark Stein, MD, Principal Investigator — Columbia University
Locations (23):
- United States (23):
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Rocky Mountain Cancer Centers USOR, Aurora, Colorado
  - Moffitt Cancer Cancer, Tampa, Florida
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Chesapeake Urology Research Associates, Towson, Maryland
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - XCancer/GU Research Network, Omaha, Nebraska
  - Rutgers Cancer Institute, New Brunswick, New Jersey
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - NYU Langone Health, Laura & Isaac Perlmutter Cancer Center, New York, New York
  - Columbia University Irving Cancer Center, New York, New York
  - UNC North Carolina Comprehensive Cancer Care Center, Chapel Hill, North Carolina
  - Duke Cancer Center, Durham, North Carolina
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - OHSU Knight Cancer Institute, Portland, Oregon
  - UT Southwestern Medical Center, Dallas, Texas
  - Virginia Cancer Specialists USOR, Fairfax, Virginia
  - Virginia Oncology Associates USOR, Norfolk, Virginia
  - Oncology and Hematology Associates Of Southwest Virginia USOR, Norton, Virginia
  - UW Carbone Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No